CLINICAL TRIAL: NCT03874728
Title: Preventing Falls in Older People Using an Innovative Connected Shoe: Development & Biomechanics Study.
Brief Title: The Effects of Minimal Shoes in Older People at Risk of Falls: The Feetback Shoe Study
Acronym: FSS
Status: Completed | Type: Observational
Sponsor: University of Liverpool (Other)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Tomasz Cudejko, Study coordinator, University of Liverpool
Other Study IDs: 4151
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Falls; Aging
Keywords: Falls; Gait; Stability; Muscle activity; Footwear; Minimal shoes; Smart shoe insoles
MeSH Terms: interventions — Community Health Workers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older people at risk of falls: Older people at risk of falls
  Interventions: Other: Minimal shoes; Other: Standardised conventional shoes; Other: Barefoot; Other: "Smart" shoe insoles

INTERVENTIONS:
Other: Minimal shoes — A minimal shoe (Vivobarefoot Ltd., London, UK) will be used.
Other: Standardised conventional shoes — The Go Walk 4.0-Pursuit shoe for women (Skechers USA, Inc.) and the Superior 2.0-Jeveno shoe for men (Skechers USA, Inc) will be used.
Other: Barefoot — Participants will conduct the assessments barefoot.
Other: "Smart" shoe insoles — Arion pressure-measuring insoles (Eindhoven, The Netherlands) will be used in the study.

SUMMARY:
A third of people over 65, and half of people over 80, fall at least once a year. Falls are the most common cause of death from injury in the over 65s and result in a significant financial burden on the whole society. Shoes directly influence balance, gait, and the subsequent risk of slips, trips and falls by altering somatosensory feedback to the foot and ankle. Minimal shoes, that is shoes lacking a firm heel cup, a rigid sole or longitudinal arch support, have shown advantages in strengthening muscles and improving balance as compared to conventional shoes. However, limited research has studied the effect of minimal shoe in older people at risk of falls. The aim of the project will be to assess the effects of minimal shoes in older people at risk of falls, compared to conventional shoes and barefoot.

DETAILED DESCRIPTION:
Study participants will attend a one-day testing session at the Movement Laboratory, University of Liverpool. Participants will be subjected to several standing and walking tests while wearing three types of footwear in a randomised order: (i) a minimal shoe, (ii) a conventional shoe, and (iii) barefoot. Participants' physical function, stability during standing and walking and an activity of lower leg muscles will be assessed in each of those three footwear conditions. Participants will also be asked about perceptions of footwear, regarding a minimal shoe and a conventional shoe. At the end of assessments, participants will be asked to complete several walking bouts while wearing a minimal shoe with "smart" shoe insoles, to determine "smart" insoles' validity in obtaining gait characteristics against a gold standard measure. Finally, those participants who volunteer to take part in a two-week follow-up study, will be asked to wear the minimal shoes with "smart" insoles during daily life for two weeks, After two weeks, they will be asked to fill in an online questionnaire asking them about total time they used the minimal shoes and insoles and about how satisfied they were with them.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 60 years old
* One of the vulnerability criteria for risk falls:

  (i) ≥ 1 self-reported falls after the age of 60; (ii) balance impairment as indicated by a score <45 on the Berg Balance Scale, by a score >2 on the simplified Tinetti Gait & Balance test or via any other validated and reliable clinical instrument used at the recruitment site; (iii) one or two criteria for physical frailty

Exclusion Criteria:

* Macro-vascular symptoms (angina, stroke or a peripheral vascular disease)
* Neuromuscular diseases (Multiple Sclerosis, Alzheimer Disease or Parkinson Disease)
* Diabetes
* Use of a walking aid (cane or walker)
* Ankle, knee, hip surgery ≤ 3 months
* Pain in the lower extremities of ≥ 8 on the numeric rating scale

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community-dwelling older adults
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go test | First day of joining the study
  Time (in seconds) to complete the Timed Up and Go test
Star Excursion Balance Test | First day of joining the study
  Reach (in centimetres) to achieve during the Star Excursion Balance Test
Postural stability | First day of joining the study
  Anterior-Posterior and latero-medial movement (in centimetres) of the centre of pressure
Dynamic stability | First day of joining the study
  Variability (standard deviations) of spatio-temporal gait characteristics
Muscle activity | First day of joining the study
  Electromyography activity for selected lower leg muscles and expressed in millivolts
Perceived attractiveness | First day of joining the study
  Scored on a 100-millimetres (mm) visual analogue scale with 0 mm being "extremely unattractive" and 100 mm being "extremely attractive"
Perceived attractiveness for others | First day of joining the study
  Scored on a 100-millimetres (mm) visual analogue scale with 0 mm being "extremely unattractive for others" and 100 mm being "extremely attractive for others"
Perceived comfort | First day of joining the study
  Scored on a 100-millimetres (mm) visual analogue scale with 0 mm being "extremely uncomfortable" and 100 mm being "extremely comfortable"
Perceived weight | First day of joining the study
  Scored on a 100-millimetres (mm) visual analogue scale with 0 mm being "extremely light" and 100 mm being "extremely heavy"
Perceived fit | First day of joining the study
  Scored on a 100-millimetres (mm) visual analogue scale with 0 mm being "poorest fit possible" and 100 mm being "best fit possible"
Perceived ease of use | First day of joining the study
  Scored on a 100-millimetres (mm) visual analogue scale with 0 mm being "most difficult as possible" and 100 mm being "as easy as imaginable"
Perceived stability | First day of joining the study
  Scored on a 100-millimetres (mm) visual analogue scale with 0 mm being "extremely unstable" and 100 mm being "extremely stable"

SECONDARY OUTCOMES:
Validity of "smart" shoe insoles | First day of joining the study
  Validity of Arion insoles against Qualisys Motion Capture System
Adherence to wearing minimal shoes in daily life | The assessment will be performed at 2 weeks
  Adherence to wearing minimal shoes with "smart" shoe insoles assessed with an online questionnaire and expressed in total time in days and hours
Satisfaction of wearing minimal shoes in daily life | The assessment will be performed at 2 weeks
  Satisfaction of wearing minimal shoes with "smart" shoe insoles assessed with an online questionnaire and expressed on a 5-point Likert scale, with the following levels: 1 - Very dissatisfied, 2 - dissatisfied, 3 - unsure, 4 - satisfied, 5 - Very satisfied.
Gait characteristics during daily life | The assessment will be performed at 2 weeks
  Gait characteristics, assessed with "smart" shoe insoles, during activities of daily life and expressed in spatio-temporal metrics

CONTACTS AND LOCATIONS:
Overall Officials: Kristiaan D'Août, PhD, Principal Investigator — University of Liverpool
Locations (1):
- University of Liverpool, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided